CLINICAL TRIAL: NCT04096443
Title: A Pilot Study of Oral FMT (Fecal Microbial Transplant) in Subjects with Multiple Sclerosis
Brief Title: Oral FMT (Fecal Microbial Transplant) in Subjects with Multiple Sclerosis
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: Yale-Griffin Prevention Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-09
Record Dates: First submitted 2019-08-07; First posted 2019-09-19 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
Keywords: Fecal microbial transplant; FMT; Pilot study
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Pre/post pilot investigational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Fecal microbial transplant capsules
  Interventions: Biological: Fecal microbial transplant (FMT)

INTERVENTIONS:
Biological: Fecal microbial transplant (FMT) — Oral fecal microbial transplant capsules

SUMMARY:
The goal of this pilot study is to determine whether fecal microbial transplant (FMT) has the potential to be an effective, safe and tolerable therapy for the treatment of multiple sclerosis (MS). The investigators plan to gather preliminary data in a small cohort of 10 to 15 adults with MS.

DETAILED DESCRIPTION:
The specific aims are to:

1. Determine the tolerability of a single dose of 30 capsules in a group of adults with MS
2. Determine whether any unexpected outcomes arise in participants who successfully complete an FMT procedure consisting of a single dose of 30 capsules
3. Determine whether successfully completed FMT leads to engraftment of donor microbiome in participants
4. If the FMT leads to engraftment of donor microbiome in participants, determine whether participants revert back to previous microbiome profiles, and if so, at what time point
5. Determine whether engrafted species following the FMT, if detected, result in any changes in immune or metabolomic parameters relative to baseline
6. Determine whether the FMT has any adverse impact, relative to baseline, on study participants' self-reported levels of fatigue, mental well-being, and health-related qualify of life
7. Determine whether the FMT has any adverse impact, relative to baseline, on study participants' neurological status, relative to baseline

The study population will consist of adults with clinically definite MS who are currently untreated with any disease-modifying therapy or are being treated with glatiramer acetate or interferon beta. The research team will offer study participants a single FMT procedure in the form of 30 oral capsules which contain fecal material. Study participants will visit Griffin Hospital facilities 8 times. The first visit will involve a clinical screening. Of the 7 remaining visits, 6 will involve data collection and one will involve the FMT procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of clinically definite multiple sclerosis (CDMS) by 2017 McDonald Criteria
2. Ages between 18 and 55 years, inclusive;
3. Expanded Disability Status Score (EDSS) between 1.0 and 6.5.
4. Currently untreated with any disease-modifying therapy (DMT) or currently being treated with glatiramer acetate or interferon beta.
5. Ability to travel to Griffin Hospital for 8 visits over a 5-month period

Exclusion Criteria:

1. Inability to give consent;
2. Non-fluency in English;
3. Inability to adhere to the protocol;
4. Inability (e.g., dysphagia) to or unwillingness to swallow capsules;
5. Active gastrointestinal infection at the time of enrollment;
6. Use of antibiotics or corticosteroids within three months of study entry;
7. Requiring or anticipating antibiotic use during the four weeks after study entry;
8. MS relapse within one month of study entry;
9. Previous use of any of the following FDA-approved disease-modifying drugs within 12 months of study entry, including natalizumab, fingolimod, siponimod, ozanimod, teriflunomide, diroximel, ocrelizumab, ofatumumab, and/or dimethyl fumarate; or any of the following off-label therapies, including rituximab and cyclophosphamide;
10. Any previous use of the following FDA-approved DMTs, including mitoxantrone, alemtuzumab, and cladribine;
11. IV immunoglobulin or plasma exchange within six months prior to study entry;
12. Known or suspected toxic megacolon and/or known small bowel ileus;
13. Major gastrointestinal surgery (e.g., significant bowel resection) within 3 months prior to enrollment (this does not include appendectomy or cholecystectomy);
14. History of total colectomy or bariatric surgery;
15. Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for active malignancy;
16. Anticipated life expectancy of less than six months;
17. Concomitant other known autoimmune diseases;
18. Concomitant pulmonary, cardiac, gastrointestinal (except as noted above) (Crohns, Colitis, inflammatory bowel, intestinal blockage), hepatic, dermatological or genitourinary disease.
19. Moderate to severe dysphagia;
20. History of alcohol abuse, as defined by the following criteria:

    Men: 5 or more alcoholic beverages per session or day, or 15 or more per week; Women: 4 or more alcoholic beverages per session or day, or 8 or more per week;
21. History of illicit drug abuse, e.g., of cocaine, heroin, PCP, and/or narcotic substances;
22. Grade 1 or greater lymphopenia, as measured at baseline/clinical screening;
23. Liver Function Tests (LFTs) greater than 1½ times upper limits of normal, as measured at baseline/clinical screening;
24. History of use of FMT or microbiome-based products (excluding probiotics) at any time, excluding this study;
25. History of severe anaphylactic or anaphylactoid food allergy;
26. History of solid organ transplantation;
27. Risk for Cytomegalovirus (CMV) or Epstein Barr virus (EBV) associated disease (at investigator's discretion, e.g., immunocompromised and negative (immunoglobulin gamma) IgG testing for CMV or EBV);
28. Women who are pregnant, lactating, planning to become pregnant, and/or not using an effective method of contraception (women of childbearing potential will undergo a pregnancy test, and will be excluded from the study if results are positive);
29. Any allergies to neomycin or similar antibiotics such as amikacin (Amikin), gentamicin (Garamycin), kanamycin (Kantrex), paromomycin (Humatin, Paromycin), streptomycin, or tobramycin (Nebcin, Tobi);
30. Any condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the study results.
31. Household contacts, including children under the age of 5 years, pregnant women, any person with an immunocompromised condition or on medications causing immunosuppression or persons 70 years or older;
32. Failure to document a COVID-19 vaccine series at least two weeks prior to study entry.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in engraftment of donor microbiome in stool samples | Pre-FMT and 4 time points post-FMT (3-7 days, 10-15 days, 40-45 days, 100-110 days)
  Evidence of engraftment as measured by 16s rRNA microbiome sequencing

SECONDARY OUTCOMES:
Change in immune markers in blood samples assessed using assays of lymphocyte phenotyping and intracellular cytokines | Pre-FMT and 2 time points post-FMT (40-45 days, 100-110 days)
  Phenotyping will be performed: for T cells - TCRβ, TCRγ, CD4, CD8, CD25, CD44, CD62L, CD69, PD1, CTLA4; for B cells - B220, CD19, CD21, CD23, CD1d, CD5, IgA, IgG1, IgG2a(c), IgG2b; for DCs - CD11c, CD11b, BDCA1, CD8, CD103, CD205 and CD86. The intracellular cytokine (ICC) panel will be IL-6, IL-10, IL-12, IL-17, TNFα, and IFNγ.
Change in neurological status using Kurtzke Functional Systems Scale (FSS) | Pre-FMT and 4 time points post-FMT (3-7 days, 10-15 days, 40-45 days, 100-110 days)
  The FSS uses a set of single-item ordinal clinical rating scales to rate levels of function in seven domains (pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, and cerebral/mental). Each single item scale ranges from 0 to 5 or 6 (0 = "normal;" 5 or 6 represents the worst level of function; and 9 = "unknown"). For each single item scale, scores representing the highest level of function are as follows: pyramidal: 6 = "quadriplegia"; cerebellar: 5 = "unable to perform coordinated movements due to ataxia"; brainstem: 5 = "inability to swallow or speak"; sensory: 6 = "sensation essentially lost below the head"; bowel and bladder: 6 = loss of bowel and bladder function"; visual: 6 = "grade 5 plus maximal visual acuity of better eye of 20/60 or less"; cerebral/mental: 5 = "dementia or chronic brain syndrome - severe or incompetent." The ratings are used in conjunction with observations and information concerning gait and use of assistive devices to rate the EDSS.
Change in neurological status using Kurtzke Expanded Disability Status Scale (EDSS) | Pre-FMT and 4 time points post-FMT (3-7 days, 10-15 days, 40-45 days, 100-110 days)
  The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10 (death due to MS) in half-point increments.
Change in self-reported health-related quality of life assessed using the Health Status Questionnaire Short-Form 36 (SF-36) | Pre-FMT and 3 time points post-FMT (10-15 days, 40-45 days, 100-110 days)
  The SF-35 has 36 questions. It has a single item covering change in health status over the last year and 8 multi-item scales. The scoring system is relatively complex and generates 8 subscales and 2 summary scores. The 8 subscales are: physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role-limitations due to emotional problems, and mental health. Two summary scales (Physical and Mental) have been derived using factor analytic methods. Scales are set up so that a higher score indicates better health. To achieve this, responses on 10 items are recoded before being added to other items on the same scale. Raw scale scores are then transformed to a 0-100 scale.
Change in self-reported mental health status assessed using Mental Health Inventory (MHI) | Pre-FMT and 3 time points post-FMT (10-15 days, 40-45 days, 100-110 days)
  The MHI consists of 18 items and assesses several domains of mental health. The scoring system generates 4 subscale scores (Anxiety, Depression, Behavioral Control, and Positive Affect) and 1 total score. The subscale and total scores range from 0-100, with higher scores indicating better mental health.
Change in self-reported levels of fatigue assessed using Modified Fatigue Impact Scale (MFIS) | Pre-FMT and 3 time points post-FMT (10-15 days, 40-45 days, 100-110 days)
  The MFIS provides an assessment of the effects of fatigue on physical, cognitive, and psychosocial function. It consists of 21 items. The items be aggregated into 3 subscales (Physical, Cognitive, and Psychosocial), as well as into a total MFIS score. All items are scaled so that higher scores indicate a greater impact of fatigue on a patient's activities. The physical subscale can range from 0-36. The cognitive subscale can range from 0-40. The psychosocialsub scale can range from 0-8. The Total MFIS score can range from 0-84.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day of FMT procedure and 5 time points post-FMT (1 day, 3-7 days, 10-15 days, 40-45 days, 100-110 days), or any time the study team is contacted by subjects who report adverse side effects
  Measured by subject's ability to consume capsules as directed without vomiting or adverse side effects (as opposed to mild side effects)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Guarnaccia, MD, Principal Investigator — Griffin Hospital; Frederick Browne, MD, Principal Investigator — Griffin Hospital
Locations (1):
- Griffin Hospital, Derby, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No